CLINICAL TRIAL: NCT02880046
Title: Study of Polyfunctionality of Anti-tumor T Lymphocytes in Cancerology: Potential Biomarker for Emerging Immunotherapies
Acronym: POLYTCANCER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: REGLOR2016/POLYT-DECARVALHO/MS
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Cancer
Keywords: immune response; T lymphocyte; PD-1/PDL-1 pathway
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Frozen PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Melanoma (LyteloMel)
- Lung cancer (TeloCap)
- Renal carcinoma (EMIR)

SUMMARY:
Purposes of this study are :

* Characterization of polyfunctionality of anti-tumor T lymphocytes using in vitro inhibition of PD-1/PDL-1 pathway
* Study and comparison of polyfunctionality of anti-tumor T lymphocytes in cohorts of patients with melanoma, lung cancer and renal carcinoma. This cancers are chosen because of use of anti-PD-1 or anti-PDL-1 antibodies
* Comparison of this technique with IFN-γ Elispot assay for detection and quantification of anti-tumor T lymphocytes after in vitro blockade of PD-1/PDL-1 pathway.

DETAILED DESCRIPTION:
In this study an immunomonitoring of specific responses of T lymphocytes to tumor-associated antigens based on detection of intracellular cytokines through flow cytometry, after stimulation with all-tumor antigens and blockade of PD-1/PDL-1 interaction is used. Peripheral blood mononuclear cells of patients with cancers are stimulated with 4 telomerase-peptides or peptides overlapping the entire sequence of survivin.

This project studies the frequency and role of polyfunctionality of anti-tumor T lymphocytes in cancerology with an in vitro technique detecting polyfunctional T lymphocytes with a better sensitivity based on removal of an inhibitory PD-1/PDL-1 pathway. It is a flow cytometry protocol with various theoretical advantages in terms of reproducibility and dynamic monitoring of functionality of different sub-populations of polyfunctional anti-tumor T lymphocytes. Moreover, it allows the study of molecular mechanisms involved in proliferation of polyfunctional anti-tumor T lymphocytes with the possibility to sort sub-populations.

The use of all-tumor antigens allows the use of this technique to evaluate the presence and prognostic or predictive value of this biomarker in various cancers.

Detection of polyfunctional anti-tumor T lymphocytes can be a biomarker of anti-tumor lymphocytic adaptive immunity and a potential eligibility or efficacy criteria for new immunotherapies, such as anti-PD-1 or anti-PDL-1 treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by melanoma (LyteloMel), lung cancer (TeloCap) or renal carcinoma (EMIR) from cohorts of medical oncology department of CHRU Besançon (France)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Frozen samples from patients affected by melanoma (LyteloMel), lung cancer (TeloCap) or renal carcinoma (EMIR) from cohorts of medical oncology department of CHRU Besançon (France).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Polyfunctionality of universal cancer peptides (UCP) and/or survivin-specific responses of T lymphocytes in presence of anti-PDL-1 antibody or isotype control, evaluated with flow cytometry | Inclusion

SECONDARY OUTCOMES:
Polyfunctionality of UCP and/or survivin-specific responses of T lymphocytes in each cohort | Inclusion
Amplitude of UCP and/or survivin-specific responses of T lymphocytes in presence of anti-PDL-1 antibody or isotype control | Inclusion
Amplitude of UCP and/or survivin-specific responses of T lymphocytes evaluated with flow cytometry or IFN-γ Elispot assay | Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo DE CARVALHO BITTENCOURT, Pr, Principal Investigator — Laboratoire d'immunologie - CHRU Nancy

IPD SHARING:
Plan to Share IPD: No